CLINICAL TRIAL: NCT06631261
Title: Comparison of Cardiopulmonary Responses to 6-Minute Stepper Test Between Individuals with Bronchiectasis and Healthy Controls
Brief Title: Cardiopulmonary Responses to 6-Minute Stepper Test in Bronchiectasis Versus Healthy Controls
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aslihan Cakmak, Principal Investigator, Hacettepe University
Other Study IDs: SBA 24/793
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Bronchiectasis Adult; Healthy Controls Group - Age and Sex-matched
Keywords: Bronchiectasis; Exercise Capacity
MeSH Terms: conditions — Bronchiectasis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Bronchiectasis: Individuals with bronchiectasis
  Interventions: Other: No intervention; Observational study
- Healthy controls
  Interventions: Other: No intervention; Observational study

INTERVENTIONS:
Other: No intervention; Observational study — No intervention

SUMMARY:
Individuals with bronchiectasis exhibit productive cough and recurrent lung infections as well as reduced exercise capacity, physical activity level, and respiratory and peripheral muscle strength. 6-minute walk test (6MWT) is often used to assess exercise capacity in chronic lung diseases. 6MWT is recommended to be performed along a flat corridor, at least 30 m long, with low pedestrian traffic, on a hard surface. To overcome technical limitations during 6MWT, 6-minute stepper test (6MST) has been proposed to assess exercise capacity. Another test that provides information about exercise capacity is the 1-minute sit-to-stand test (1STS). To our knowledge, there is limited information about different exercise tests including 6MST and 1STS and cardiopulmonary responses to these tests in individuals with bronchiectasis. Therefore, this study aims to compare the responses to the 6MST between individuals with bronchiectasis and healthy controls and to investigate the relationships among 6MST, 6MWT, and 1STS responses and muscle strength.

ELIGIBILITY:
Bronchiectasis group - Inclusion criteria for the study:

* Being 18 years of age and older,
* Having a clinically stable bronchiectasis,
* To cooperate with the tests to be performed,
* Not having a cardiovascular disease, orthopedic or neurological problem that may affect the tests,
* Being willing to participate in the study.

Bronchiectasis group - Exclusion criteria:

* Being in an acute exacerbation period,
* Having a cardiovascular, orthopedic or neurological problem that may affect the tests,
* Not being willing to participate in the study.

Control group - Inclusion criteria for the study:

* Being 18 years of age and older,
* To cooperate with the tests to be performed,
* Not having a cardiovascular, orthopedic or neurological problem that may affect the tests,
* Being willing to participate in the study.

Control group - Exclusion criteria:

- Individuals with any known internal disease and those who do not volunteer to participate in the study will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with bronchiectasis and healthy controls
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2026-01-18 (Estimated); Study Completion 2026-01-18 (Estimated)

PRIMARY OUTCOMES:
Maximal inspiratory pressure | 1st day
  Maximal inspiratory pressure (MIP) and will be measured using aa mouth-piece pressure measurement device. The measurement will be repeated three times so that there will be no difference of 10 cmH₂O or 10%, and the highest value will be used for analysis.
Maximal expiratory pressure | 1st day
  Maximal expiratory pressure (MEP) and will be measured using a mouth-piece pressure measurement device. The measurement will be repeated three times so that there will be no difference of 10 cmH₂O or 10%, and the highest value will be used for analysis.
Peripheral muscle strength | 1st day
  Peripheral muscle strength will be assessed using a portable dynamometer. The peripheral muscle strength test will be repeated three times for the right and left sides.
6-minute stepper test responses | 1st day
  6-minute stepper test will be performed, and the number of repetitions will be recorded. Cardiopulmonary responses before and after 6-minute stepper test will be recorded. 6-minute stepper test will be performed twice with 30 minutes apart.
1 minute sit-to-stand test responses | 1 minute sit-to-stand test will be performed and the repetitions will be recoded. Cardiopulmonary responses will be recorded before and after the test.
  1 minute sit-to-stand test will be performed and the repetitions will be recoded. Cardiopulmonary responses will be recorded before and after the test.
6-minute walk test responses | 1st day
  6-minute walk test will be performed, and the distance walked will be recorded. Cardiopulmonary responses before and after 6-minute walk test will be recorded.

SECONDARY OUTCOMES:
Dyspnea | 1st day
  The modified Medical Research Council (mMRC) dyspnea scale will be used for dyspnea assessment. The mMRC dyspnea scale is a scale in which individuals choose the expression that best describes their dyspnea level from among 5 expressions related to shortness of breath. The higher the degree, the more severe the shortness of breath.
Charlson Comorbidity Index | 1st day
  Charlson Comorbidity Index (CCI) will be used to query accompanying comorbidities. Higher CCI scores indicate a greater burden of comorbid conditions.
Bronchiectasis Severity Index | 1st day
  Bronchiectasis Severity Index will be used to evaluate disease severity and prognosis in bronchiectasis. It is calculated by respiratory function, age, chronic colonization with Pseudomonas aeruginosa and other bacterial infections, shortness of breath and radiological extent of the disease. Based on Bronchiectasis Severity Index, bronchiectasis severity is defined as mild (0-4), moderate (5-8) and severe (≥9).
Forced vital capacity | 1st day
  Pulmonary function test using a spirometer will be performed. Forced vital capacity will be recorded.
Forced expiratory volume in one second | 1st day
  Pulmonary function test using a spirometer will be performed. Forced expiratory volume in one second will be recorded.
Forced expiratory volume in one second/forced vital capacity ratio | 1st day
  Pulmonary function test using a spirometer will be performed. Forced expiratory volume in one second/forced vital capacity ratio will be recorded.
Peak expiratory flow | 1st day
  Pulmonary function test using a spirometer will be performed. Peak expiratory flow will be recorded.
Forced mid-expiratory flow (FEF25-75) | 1st day
  Pulmonary function test using a spirometer will be performed. Forced mid-expiratory flow (FEF25-75) will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No